CLINICAL TRIAL: NCT00003463
Title: Phase I Treatment of Adults With Recurrent Supratentorial High Grade Glioma With Gliadel Wafers Plus Irinotecan (CPT-11)
Brief Title: Carmustine Wafers Plus Irinotecan in Treating Patients With Recurrent Supratentorial High Grade Gliomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 0901; DUMC-0901-02-5R4; DUMC-0901-02-5R2; DUMC-000901-00-5R2; DUMC-000901-01-5R3; DUMC-0797-99-5RI; DUMC-796-98-5; DUMC-98065; UCLA-9812060; NCI-G98-1464; DUMC-0901-01-5R3; CDR0000066497 (Other: NCI)
Record Dates: First submitted 1999-11-01; First posted 2003-09-25 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-02

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult brain stem glioma; adult glioblastoma; adult anaplastic astrocytoma; adult mixed glioma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioblastoma; Astrocytoma; Glioma; Gliosarcoma | interventions — Carmustine; Irinotecan; Surgical Procedures, Operative

INTERVENTIONS:
Drug: carmustine
Drug: irinotecan hydrochloride
Drug: polifeprosan 20 with carmustine implant
Procedure: surgical procedure

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of carmustine wafers plus irinotecan in treating patients with recurrent supratentorial high grade gliomas.

DETAILED DESCRIPTION:
OBJECTIVES:

* Define the maximum tolerated dose of irinotecan given in combination with Gliadel wafers (carmustine) in patients with recurrent glioblastoma multiforme, anaplastic astrocytoma, or gliosarcoma.
* Define the toxicity of irinotecan given in combination with Gliadel wafers in these patients.

OUTLINE: This is a dose escalation study.

All patients undergo surgical resection. At the time of surgery, up to eight Gliadel wafers (containing carmustine) are implanted in the resected tumor cavity.

Cohorts of 3 patients each receive escalating doses of irinotecan IV over 90 minutes once weekly within 3 weeks after Gliadel wafer implantation. One course of treatment consists of 4 weeks of irinotecan and 2 weeks of rest. If 1 patient experiences dose limiting toxicity (DLT) at a dose level, an additional 3 patients are entered at that same dose level. If 2 patients experience DLT, the maximum tolerated dose (MTD) has been surpassed and a total of 6 patients are treated at the previous dose level. The MTD is defined as the highest dose in which no more than 1 of 6 patients experiences DLT.

Treatment continues for up to 12 courses in the absence of unacceptable toxicity and disease progression.

Patients are followed for at least 4 months.

PROJECTED ACCRUAL: Approximately 18 patients will be accrued into this study over 9 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed recurrent supratentorial glioblastoma multiforme, anaplastic astrocytoma, or gliosarcoma
* Must be able to undergo surgical resection
* At least 1 bidimensionally measurable lesion documented on Gd-MRI within 72 hours after surgical implantation of Gliadel wafers
* Not requiring immediate radiotherapy

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 70-100%

Life expectancy:

* Greater than 12 weeks

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 125,000/mm^3
* Hematocrit at least 29%

Hepatic:

* Bilirubin less than 1.5 times upper limit of normal (ULN)
* SGOT or SGPT less than 2.5 times ULN
* Alkaline phosphatase less than 2 times ULN

Renal:

* BUN less than 1.5 times ULN
* Creatinine less than 1.5 times ULN

Neurological:

* Must be neurologically stable

Other:

* HIV negative

  * No AIDS-related illness
* No nonmalignant systemic disease that would make patient a poor medical risk
* No acute infection requiring intravenous antibiotics
* Not pregnant or nursing

  * Negative pregnancy test 24 hours prior to study
* Effective contraception required of all fertile patients

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior irinotecan
* At least 6 weeks since chemotherapy unless there is unequivocal evidence of tumor progression after chemotherapy

Endocrine therapy:

* At least 1 week of nonincreasing dose of steroids prior to study

Radiotherapy:

* At least 6 weeks since radiotherapy unless there is unequivocal evidence of tumor progression after radiotherapy
* No concurrent radiotherapy

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-07; Primary Completion 2002-07 (Actual); Study Completion 2002-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry S. Friedman, MD, Study Chair — Duke Cancer Institute
Locations (2):
- United States (2):
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Duke Comprehensive Cancer Center, Durham, North Carolina